CLINICAL TRIAL: NCT00370812
Title: The Role of Amniotic Membrane Transplantation in Ocular Chemical Burns
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8528
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Eye Burns
Keywords: amniotic membrane transplantation; ocular chemical burns
MeSH Terms: conditions — Eye Burns

ARMS (2):
- A (Active Comparator): AMT with conventional medical therapy
  Interventions: Procedure: amniotic membrane transplantation
- B (Active Comparator): Medical treatment alone
  Interventions: Procedure: amniotic membrane transplantation

INTERVENTIONS:
Procedure: amniotic membrane transplantation — AMT with conventional medical therapy (group A) or medical treatment only (group B). AMT will be performed within 24h of presentation. Amniotic membrane will remain in place for 7-14 days.

SUMMARY:
This is a randomized clinical trial study to identify the role of AMT (amniotic membrane transplantation) in treating epithelial defect, symblepharon prevention preventing corneal vascularization and opacity decreasing pain and improving visual acuity, and patients with acute chemical burns.

DETAILED DESCRIPTION:
The study is on patients with grade II-IV acute ocular chemical burns (Roper - Hall classification) in the first 2 weeks of injury.

After topical anesthesia, all patients initially will receive first aid therapy; which included irrigation with normal saline to normalize ocular surface PH and removal of early particulate maeuil and debris. After complete examination and obtaining informed consent, the patients will be randomized using a treatment assignment list to either AMT with conventional medical therapy (group A) or medical treatment only (group B). In the patients with bilateral injuries the eyes will be randomized separately. AMT will be performed within 24h of presentation. amniotic membrane will remain in place for 7-14 days. The patients will be examined at days 1, 3, 7, 10, 14, 21, 28 and then biweekly until 3 months and monthly until (1 year in every visit, visual acuity (by sneillen charts), reduction of pain (subjectively) size of corneal epithelial defect (by fluorseein satiny extent of corneal vascularization and opacity, and symblepharon formation will be assessed. Digital photographs at each visit will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chemical eye burn grade 2-4
* Burning has been occurred in 2 weeks

Exclusion Criteria:

* Grade I burnings
* More than 2 weeks have passed of burning
* Follow up of the patients has been disconnected in 6 month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Days 1, 3, 7, 10, 14, 21, 28 and then every 2weeks until 3 months and monthly until 1 year
Pain | Days 1, 3, 7, 10, 14, 21, 28 and then every 2weeks until 3 months and monthly until 1 year
Symblepharon formation | Days 1, 3, 7, 10, 14, 21, 28 and then every 2weeks until 3 months and monthly until 1 year
Epithelial defect healing | Days 1, 3, 7, 10, 14, 21, 28 and then every 2weeks until 3 months and monthly until 1 year
Corneal opacity and vascularization | Days 1, 3, 7, 10, 14, 21, 28 and then every 2weeks until 3 months and monthly until 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Baradaran Raffiee, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Labbafinejad Medical Center, Tehran, Tehran Province, Iran